CLINICAL TRIAL: NCT04900740
Title: Evaluation of a Tissue Glue SecurePortIV on Prevention of Phlebitis and Migration of PICC and Midline Catheters in Adult Patients
Brief Title: Evaluation of Tissue Glue on PICC and Midline Catheters Insertion Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FNO-PICC-03; 03/RVO-FNOs/2021 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2021-05-13; First posted 2021-05-25 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Adult Patients With Mid-term or Long-term Venous Access
Keywords: peripherally inserted central catheter; midline; cyanoacrylate tissue glue; tissue glue; phlebitis; catheter migration
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: The patients will be enrolled into one of two study groups, depending on the decision of the attending physician.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care - catheter fixation with surgical stitch (Active Comparator): In patients indicated for this type of treatment, as per the attending physician, the catheter will be fixed in the standard way, using a surgical stitch.
  Interventions: Device: Catheter fixation with surgical stitch
- Experimental - catheter fixation with glue (Experimental): In patients indicated for this type of treatment, as per the attending physician, the catheter will be fixed using the glue.
  Interventions: Device: Catheter fixation with glue (cyanoacrylate tissue glue Secure PortIV)

INTERVENTIONS:
Device: Catheter fixation with surgical stitch — The catheter will be fixed using the standard procedure - surgical stitch.
  Arms: Standard care - catheter fixation with surgical stitch
Device: Catheter fixation with glue (cyanoacrylate tissue glue Secure PortIV) — The catheter will be fixed using the experimental procedure - novel surgical glue.
  Arms: Experimental - catheter fixation with glue

SUMMARY:
The study will evaluate a new type of cyanoacrylate tissue glue Secure PortIV on the insertion site of the PICC (Peripherally inserted central catheter) or Midline catheters. Fixation of the catheter with the tissue glue should prevent incidents of mechanical and infective phlebitis as well as external migrations of the catheters.

DETAILED DESCRIPTION:
In the study, 125 subjects will receive the new tissue glue Secure PortIV and 125 subjects will be provided standard care. The tissue glue will be applied immediately after insertion. Evaluation and re-evaluation of the site will be done on the first and seventh day after insertion using VIP and CLISA (Central-Line Insertion Site Assessment) scale and on the seventh day with taking a swab from the insertion site; the external length will be measured on the first and the seventh day, in order to observe the migration or not.

The goal of the study is to evaluate the benefits of the cyanoacrylate tissue glue Secure PortIV in the prevention of mechanical and infective phlebitis and external migration of the catheter.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* need of long-term venous access
* consent with participation in the study

Exclusion Criteria:

* pediatric population
* not signing the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of mechanical and infective phlebitis | Up to 6 months
  The incidence of mechanical and infective phlebitis will be measured in the group with the cyanoacrylate tissue glue in comparison with the standard treatment

SECONDARY OUTCOMES:
The incidence of external migration of the catheter | Up to 6 months
  The incidence of external migration of the catheter will be measured in the group with the cyanoacrylate tissue glue in comparison with the standard treatment

CONTACTS AND LOCATIONS:
Overall Officials: Iveta Constantine, Bc., MSc., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Scoppettuolo G, Dolcetti L, Emoli A, La Greca A, Biasucci DG, Pittiruti M. Further benefits of cyanoacrylate glue for central venous catheterisation. Anaesthesia. 2015 Jun;70(6):758. doi: 10.1111/anae.13105. No abstract available. PMID 25959189
- [Background] Di Puccio F, Giacomarro D, Mattei L, Pittiruti M, Scoppettuolo G. Experimental study on the chemico-physical interaction between a two-component cyanoacrylate glue and the material of PICCs. J Vasc Access. 2018 Jan;19(1):58-62. doi: 10.5301/jva.5000816. PMID 29148010
- [Background] Seckold T, Walker S, Dwyer T. A comparison of silicone and polyurethane PICC lines and postinsertion complication rates: a systematic review. J Vasc Access. 2015 May-Jun;16(3):167-77. doi: 10.5301/jva.5000330. Epub 2015 Jan 23. PMID 25634150
- [Background] Gorski LA, Hadaway L, Hagle ME, Broadhurst D, Clare S, Kleidon T, Meyer BM, Nickel B, Rowley S, Sharpe E, Alexander M. Infusion Therapy Standards of Practice, 8th Edition. J Infus Nurs. 2021 Jan-Feb 01;44(1S Suppl 1):S1-S224. doi: 10.1097/NAN.0000000000000396. No abstract available. PMID 33394637
- [Background] Di Giacomo M. Comparison of three peripherally-inserted central catheters: pilot study. Br J Nurs. 2009 Jan 8-21;18(1):8-16. doi: 10.12968/bjon.2009.18.1.32071. PMID 19127226 (Retraction: PMID 24930146 Br J Nurs. 2014 May 8-21;23(9):S25)
- [Background] Igarashi A, Okuno T, Shimizu T, Ohta G, Ohshima Y. Mechanical stimulation is a risk factor for phlebitis associated with peripherally inserted central venous catheter in neonates. Pediatr Int. 2021 May;63(5):561-564. doi: 10.1111/ped.14476. Epub 2021 May 7. PMID 32964580
- [Background] Walshe LJ, Malak SF, Eagan J, Sepkowitz KA. Complication rates among cancer patients with peripherally inserted central catheters. J Clin Oncol. 2002 Aug 1;20(15):3276-81. doi: 10.1200/JCO.2002.11.135. PMID 12149302
- [Background] Pinelli F, Balsorano P, Mura B, Pittiruti M. Reconsidering the GAVeCeLT Consensus on catheter-related thrombosis, 13 years later. J Vasc Access. 2021 Jul;22(4):501-508. doi: 10.1177/1129729820947594. Epub 2020 Aug 8. PMID 32772785